CLINICAL TRIAL: NCT06652880
Title: Exploring the Preliminary Effects of a Digital Parenting and Recovery Support Intervention for Pregnant People Seeking Recovery from Opioid Use Disorders: a Pilot Randomized Control Trial
Brief Title: Digital Support Intervention for Pregnant People with Opioid Use Disorders
Acronym: PARENTSS
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Phyllis Raynor, Clinical Assistant Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pro00136341
Record Dates: First submitted 2024-09-16; First posted 2024-10-22 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2024-09

CONDITIONS: Digital Intervention; Bibliotherapy
Keywords: PARENTSS project; Opioid Use Disorders; Pregnancy; Postpartum; Methadone; Buprenorphine; Digital technology; digital apps
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Bibliotherapy

STUDY DESIGN:
Intervention Model Description: The intervention is access to a digital application that provides parenting and recovery support on the participant's smartphone.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Customized Digital Application group (Intervention) (Experimental): Participants are assigned to one of two groups where they will receive one type of parenting support. The intervention group will receive a smartphone app which provides access to comprehensive resources related to parenting and recovery.
  The intervention group will be observed to determine how frequently they use the digital app, thoughts about it, and what was found to be helpful. This will occur over a 12-week period.
  The intervention group will complete surveys over the study period through the digital app. The times for survey completion are within one week after agreeing to participate in the study, after 6 weeks, and 12 weeks. The surveys include questions about personal history, drug usage and cravings, missed follow-up medical appointments, and parenting outcomes. An interview with the PI at 12 weeks post-delivery.
  Interventions: Device: Digital technology
- Parenting book as support for control group (Active Comparator): The bibliotherapy control group will receive a book on what to expect as a parent the first year after delivery.
  The control group will complete surveys over the study period and are given the option to complete surveys by phone or videoconference with a Team member. The times for survey completion are within one week after agreeing to participate in the study, after 6 weeks, and 12 weeks. The surveys include questions about personal history, drug usage and cravings, missed follow-up medical appointments, and parenting outcomes. An interview with the PI at 12 weeks post-delivery.
  Interventions: Other: Bibliotherapy

INTERVENTIONS:
Device: Digital technology — The digital app is a customized comprehensive self-management platform designed to provide recovery and parenting support for individuals with substance use disorders.
  Other Names: digital app
  Arms: Customized Digital Application group (Intervention)
Other: Bibliotherapy — Bibliotherapy control group will receive parenting book what to expect the first year.
  Other Names: book
  Arms: Parenting book as support for control group

SUMMARY:
The goal of this pilot randomized feasibility study is to explore the benefits of providing parenting and recovery support for pregnant people with Opioid Use Disorders through digital technology (e.g. smartphones). The main question it aims to answer is:

• What is the feasibility of providing customized digital parenting and recovery supports to pregnant people with Opioid Use Disorders residing in natural communities?

o Feasibility data includes data on study interest, eligibility, time to enroll, participant training on digital app usage, attrition;

Secondary outcome exploratory data will include MOUD treatment retention, missed follow up prenatal and early postpartum appointments, drug usage, and parenting outcomes (i.e., scores on the Parental sense of competency scale, Self-rated abilities for health practices scale, and Self-efficacy in infant care scale) through self-report; The intervention group only will also be observed regarding app usage, frequency of use, resources accessed, thoughts about the app, and what was found to be helpful.

Researchers will compare the bibliotherapy control group to determine clinical differences in secondary outcomes.

Participants will complete the following tasks:

* Schedule an online meeting with the research team to receive more information about the study. Once consented to participate, the participant will be randomly assigned to one of the groups.
* Complete survey questions within one week after agreeing to participate in the study, after 6 weeks, and 12 weeks. The surveys include questions about drug usage, missed follow-up medical appointments, and parenting outcomes. The total time to complete the survey after consenting to be in the study will take approximately 40 minutes. The total time to complete the surveys after the six week and 12-week study period should take no more than 30 minutes.
* Complete a one-hour virtual interview at three months post-delivery (by phone or computer) about the study experience.

ELIGIBILITY:
Inclusion Criteria:

Female, pregnant, greater 13 weeks gestational age

* Opioid Dominant Use Disorder and Primary Phenotype
* Residing in natural home environment
* minimum of 18 years of age
* Able to speak and understand English
* Able to understand and provide informed consent

Exclusion Criteria:

* Not pregnant, has active illicit opioid use and not currently in treatment
* a violent criminal history
* cannot read and communicate in English

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-06-04 (Actual); Primary Completion 2025-08-28 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment and Retention: Number of communications regarding study interest, number of interested persons eligible/ineligible, No. of study refusals; study attrition rates | 12 week study period; final data collection (qualitative interview) at 3 months post-delivery
  Recruitment - recruitment measures (e.g., total time, direct calls regarding interest, number eligible/ineligible, refusals) (Qualitative) Qualitative data via interviews at the end of the study period with each participant in the Intervention group regarding type of smart phone used/model; overall experience using the app, times and situations when participants were more likely to use app as a resource, app features most helpful in supporting recovery from OUD, app features most helpful in supporting parenting, and preferences regarding initiation of intervention. Attrition data --duration of time that individuals engaged with the app; participated in the study

SECONDARY OUTCOMES:
Treatment retention: Qualitative interview 3 months post delivery: responses to questions regarding status in treatment for Opioid Use Disorder, attendance to postpartum appointments, scheduled baby visits. | Qualitative interview at 3 months post-delivery
  Participants will be asked to participate in an interview at 3 months post-delivery with a research team member. Information regarding medical appointments will be collected.
Recovery Capital: Quantitative measure: Total scores on the Brief Assessment of Recovery Capital scale. | 12 week study period; final data collection (qualitative interview) at 3 months post-delivery
  Participants will be asked to complete the Brief Assessment of Recovery Capital (BARC-10) scale at certain timepoints during the 12 week study period, at the end of the 12 week study period and at 3 months post-delivery. Brief Recovery capital scale is designed to evaluate a person's resources and strengths (i.e., recovery capital) that can support their recovery from substance use disorders. Participants rate their agreement with each statement in the BARC-10 from "Strongly Disagree" (with a value of 1) to "Strongly Agree" (with a value of 6). The score for each question is added together to create the participant's total score. Total scores can range from 10 to 60, with higher scores indicating greater recovery capital.
Parenting outcomes: Quantitative measures: Total scores on the self-rated abilities for health practices scale (SRAHP) | 12 week study period
  Participants will be asked to complete surveys at baseline, 6 weeks and at 12 weeks. The SRAHP is a 28-item, 5-point scale to measure self-perceived ability to implement health-promoting behaviors. SRAHP contains four subscales. Items are rated from 0 (not at all) to 4 (completely). Total scores range from 0-112. Higher scores indicate greater self-efficacy.
Parenting outcomes: Quantitative measures: Total scores on the parental sense of competence scale (PSOC) | 12 week study period
  Participants will be asked to complete surveys at baseline, 6 weeks and at 12 weeks. The PSOC is a self-report measure that aims to assess one's perceived efficacy and satisfaction with parenting. The PSOC is a 17 item scale, with 2 subscales. Each item is rated on a 6-point Likert scale anchored by 1 = "Strongly Disagree" and 6 = "Strongly Agree". A higher score indicates a higher parenting sense of competency.
Parenting outcomes: Quantitative measures: Total scores on the self-efficacy in infant care scale (SICS) | 12 week study period
  Participants will be asked to complete surveys at baseline, 6 weeks and at 12 weeks. SICS is a 44 item questionnaire s a self-administered to assess maternal judgments about the ability to care for the baby during the first year of life. Each item is rated on a 5 point Likert scale anchored by 1 = "strongly disagree" and 6 = "strongly agree". Higher scores indicate higher self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Phyllis A Raynor, PHD, Principal Investigator — University of South Carolina
Locations (1):
- MUSC Health Institute of Psychiatry, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No
primary feasibility outcome data and secondary treatment retention data will be shared in aggregate to protect participant confidentiality.